CLINICAL TRIAL: NCT06760767
Title: Investigation of The Effectiveness of Pelvic Floor Physiotherapy Combined With Sexual Therapy in Vaginismus Treatment
Brief Title: Pelvic Floor Physiotherapy Combined With Sexual Therapy in Vaginismus Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Gülay Aras, Principal investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-222
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Women Health; Physiotherapy; Exercise
Keywords: Sexual Dysfunction; Sexual Therapy; Electromyography; Pelvic Floor Physiotherapy; Vaginismus
MeSH Terms: conditions — Motor Activity; Sexual Dysfunction, Physiological; Vaginismus

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group received pelvic floor physiotherapy combined with sexual therapy twice a week for 6 weeks.
  Interventions: Behavioral: sexual therapy; Behavioral: Pelvic floor physiotherapy combined with sexual therapy
- Control Group (Experimental): Participants in the control group received sexual therapy twice a week for 6 weeks.
  Interventions: Behavioral: sexual therapy

INTERVENTIONS:
Behavioral: sexual therapy — In sexual therapy sessions, sexual education, cognitive restructuring, body awareness exercises, systematic desensitization, relaxation training, individual and partner home exercise training and dilator treatment were applied with the supervision of a physiotherapist. All techniques and stages were not applied in the same session and were used with a certain progression
Behavioral: Pelvic floor physiotherapy combined with sexual therapy — Pelvic floor physiotherapy combined with sexual therapy was applied in the experimental group. Sexual therapy techniques were added appropriately before, during and after the pelvic floor physiotherapy session. In the pelvic floor physiotherapy sessions, pelvic floor muscle training, biofeedback, electrotherapy, manual therapy applications, breathing exercises, stretching and relaxation exercises were applied with the physiotherapist. Pelvic floor physiotherapy techniques and stages were applied in the same session and followed a certain progression.
  Arms: Intervention Group

SUMMARY:
Studies on pelvic floor physiotherapy in individuals diagnosed with vaginismus are quite limited in the literature. While current studies have focused on certain physiotherapy modalities, the literature is quite limited in terms of combined rehabilitation programs. There is a need for non-invasive therapy methods that can be an alternative for the patient and client population whose vaginismus problem continues after behavioral therapies. No studies on pelvic floor physiotherapy combined with sexual therapy have been found in the literature. In this context, our study aimed to examine the effectiveness of pelvic floor physiotherapy combined with sexual therapy in individuals diagnosed with vaginismus.

DETAILED DESCRIPTION:
Vaginismus is a sexual dysfunction defined as recurrent or persistent difficulty or impossibility of sexual intercourse due to involuntary contractions of the muscles in the vaginal area in women. This condition is usually associated with excessive tension and spasm of the pelvic floor muscles and adductor muscles when evaluated in terms of these muscle groups.

Sexuual therapy includes the placement of dilators of graduated sizes by the therapist at home or in a clinical setting, guided by both the patient and the partner, for systematic desensitization to vaginal penetration, and sexual education to alleviate the psychological impact of the condition. This method is most frequently used in studies and the reported success rates are quite high.

Various techniques such as breathing and relaxation exercises, local tissue desensitization, vaginal dilators, biofeedback and manual therapy are used within the scope of pelvic floor physiotherapy in the treatment of vaginismus. There are studies in the literature investigating the effectiveness of biofeedback exercises in the treatment of vaginismus with a 100% success rate. It has also been reported that the combined application of pelvic floor exercises with behavioral sexual therapy provides significant improvement. In this study aimed to examine the effectiveness of pelvic floor physiotherapy combined with sexual therapy in individuals diagnosed with vaginismus.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with vaginismus,
* Being between the ages of 20-45,
* Having an active sexual partner in the last 6 months,
* Not being in the accompanying physiotherapy or psychotherapy process.

Exclusion Criteria:

* Diagnosed with or treated for vulvodynia and/or vulvar vestibulitis,
* Having a pacemaker,
* Not being able to give personal consent,
* Having a physical problem that would prevent treatment.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Surface Electromyography (sEMG) | 0-6 weeks
  A 2-channel Neurotrac MyoPlus 4 Pro (Verity Medical, UK) surface electromyography (sEMG) device with testing and biofeedback features was used to measure the activity of the pelvic floor muscles, adductor and muscles

SECONDARY OUTCOMES:
Female Sexual Function Index (FSFI) | 0-6 weeks
  The FSFI consists of 19 questions and aims to determine the ongoing sexual functions of the person in the last four weeks.
The Vaginal Penetration Cognition Questionnare (VPCQ) | 0-6 weeks
  The questions in this questionnaire are aimed at investigating thoughts related to vaginal penetration.
"Does sexual intercourse occur?" | 0-6 weeks
  Before and after the treatment, the participants were asked the question "Does sexual intercourse occur?" and their answers were collected as "Yes" and "No".

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Aras Bayram, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)